CLINICAL TRIAL: NCT00886301
Title: Fatty Liver and Ectopic Fat in Overweight and Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-PP-08
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Steatohepatitis
Keywords: overweight; obesity; steatohepatitis; ectopic fat
MeSH Terms: conditions — Fatty Liver; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): obese or overweight patients with fatty liver or ectopic fat
  Interventions: Procedure: liver biopsy

INTERVENTIONS:
Procedure: liver biopsy — liver biopsy

SUMMARY:
The aim of the study is to find new clinico-biological and medical imaging parameters associated with non alcoholic steatohepatitis in overweight and obese patients.

DETAILED DESCRIPTION:
Non invasive assessment of liver fibrosis and liver inflammation and steatosis is clinically relevant in patients exposed to non alcoholic fatty liver diseases.

The aim of the study is to find new clinico-biological and medical imaging parameters associated with non alcoholic steatohepatitis in overweight and obese patients.

Fatty liver and ectopic fat accumulation will be particularly assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 40
* ALAT level superior to normal level even after 3 months of diet
* alcohol consumption < 20 g/j for women and < 30 g/j for men

Exclusion Criteria:

* HIV, hepatitis B virus, hepatitis C virus positive
* known hemochromatosis
* glycemia > 1.26 g/L or under anti-diabetic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2014-10-02 (Actual); Study Completion 2014-10-02 (Actual)

PRIMARY OUTCOMES:
Liver status will be will be determined by liver biopsy, non invasive liver assessment. Biological and medical imaging parameters will be use to characterize our patients. | at inclusion and at year 1

SECONDARY OUTCOMES:
Non invasive liver assessment, biological and medical imaging parameters will be use to characterize our patients. | at year 1

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe ANTY, Dr, Principal Investigator — Hepatogastroentérology, CHU de Nice
Locations (1):
- Hepatogastroenterology, Hôpital l'Archet, CHU de Nice, Nice, France